CLINICAL TRIAL: NCT04411147
Title: A Longitudinal Study of COVID-19 Sequelae and Immunity
Status: Active, not recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200123; 20-I-0123
Record Dates: First submitted 2020-05-30; First posted 2020-06-02 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01-09

CONDITIONS: COVID-19
Keywords: Coronavirus; SARS-CoV-2; Medical Sequelae; Antibody and Cell-mediated Immune Responses; Protective Immunity; Natural History
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Close Contacts: Individuals without COVID-19 diagnosis, lived in same home as a survivor during illness, were within 6 feet of a COVID-19 case for a prolonged period of time or had direct contact with secretions
- COVID-19 Survivor: Individuals with documented prior COVID-19 infection and who have recovered

SUMMARY:
Background:

COVID-19 is a disease caused by the SARS-CoV-2 virus. It infects the respiratory tract. Some people who get COVID-19 have only mild symptoms. But for others, infection leads to pneumonia, respiratory failure, and, in some cases, death. Researchers want to learn more about any effects that may persist after people recover from COVID-19.

Objective:

To learn about any long-term medical problems that people who have recovered from COVID-19 might have, and whether they develop an immune response to SARS-CoV-2 that provides protection against reinfection.

Eligibility:

People age 18 and older who have recovered from documented COVID-19 or were in close contact with someone who had COVID-19 but did not get the infection

Design:

Participants will be screened over 2 visits. During visit 1, they will answer questions about any symptoms they are having and will be tested for SARS-CoV-2 infection which will involve a nasal swab sample or other FDA approved test. If the test is negative, they will proceed to the second visit, which will include:

Physical examination

Medical history

Mental health interview (which may be recorded if the participant agrees)

Chest x-ray (for recovered COVID-19 participants only)

Blood and urine tests

Pregnancy test (if needed)

Lung function test (for recovered COVID-19 participants only)

6-minute walk test (for recovered COVID-19 participants only)

Questionnaires about their general and mental health

Leukapheresis to collect white blood cells (optional).

Participants will be put into 1 of 2 groups: the COVID-19 group or the close contact group.

Participants will have study visits every 6 months for 3 years. They will repeat some of the screening tests. Participants in the COVID-19 group may have visits more often if they develop symptoms that suggest re-infection with SARS-CoV-2.

DETAILED DESCRIPTION:
Study Description:

This is a longitudinal cohort study to evaluate the clinical sequelae of acute COVID-19 and characterize the immune response to SARS-CoV-2. Household contacts of the COVID-19 cohort will also be recruited and serve as a control group.

Objectives:

* Characterize the medical sequalae and persistent symptoms following recovery from COVID-19 in a cohort of disease survivors.
* Estimate the incidence and risk factors for post-COVID-19 medical sequalae.
* Characterize antibody and cell-mediated immune responses to SARS-CoV- 2 in disease survivors
* Characterize evolution of the antibody and T cell-mediated responses to SARS-CoV-2 in survivors over time
* Evaluate survivors for evidence of re-infection with future waves of COVID-19 to determine if initial infection confers long-term protective immunity
* Determine the incidence of clinically silent infection in household contacts
* Characterize the mental health status of survivors and controls including medical trauma related sequelae

Endpoint:

Establish a clinically well characterized cohort of persons recovered from COVID-19 and close contacts of persons with COVID-19

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, all individuals must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study
2. Age 18 years or older.
3. Ability of participant to understand and the willingness to sign a written informed consent document.
4. Hemoglobin of 9.0 gm/dl or higher
5. Willingness to give consent for the storage of blood samples for research.
6. Have a physician or clinic outside NIH to manage underlying medical conditions or agreeing to establish care with an outside physician or clinic for any medical conditions requiring treatment that may be diagnosed as a result of protocol participation.

COVID-19 Survivor Group

1. Documented prior COVID-19 as evidenced by:

   1. detection of SARS-CoV-2 RNA or antigen in nasopharyngeal swab, sputum or other sample source with EUA/approval from the FDA; or
   2. a positive antibody test using an assay that has received emergency use authorization (EUA) from the Food and Drug Administration (FDA) and a history clinical manifestation compatible with COVID-19.
2. Greater than 6 weeks since onset of COVID-19 symptoms and no fever for at least 1 week. For individuals with asymptomatic infection, screening will not occur until at least 4 weeks after the last positive SARS-CoV-2 PCR or antigen test.

COVID-19 Close Contact

1. Living in the same household as a COVID-19 survivor during the time of illness or, being within approximately 6 feet (2 meters) of a COVID-19 case for a prolonged period of time or having direct contact with infectious secretions of a COVID-19 case (e.g., being coughed on).
2. No diagnosis of COVID-19 or current symptoms suggestive of COVID-19

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Current abuse of alcohol or other drugs that, in the judgement of the Principal Investigator (PI) could interfere with patient compliance.
2. Inability to travel to the NIH Clinical Center for study visits
3. Any medical or mental health condition that, in the judgement of the PI, would make the volunteer unable to participate in the study.
4. Positive SARS-CoV-2 PCR at screening visit
5. Positive test for antibodies to SARS-CoV-2 nucleocapsid protein at the screening visit (control group only).
6. History of any of the following in the past 14 days: fever > 38.2 degrees Celsius; new or worsening respiratory symptoms (e.g. cough, dyspnea).
7. Pregnancy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Clinical
Sampling Method: Non-Probability Sample
Enrollment: 583 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Risk Factors for Medical Sequelae in COVID-19 Survivors | Screening-Month 36
  Estimate the incidence and risk factors for post-COVID-19 medical sequalae.
Mental health status in COVID-19 survivors and contacts | Screening-Month 36
  Characterize the mental health status of survivors and controls including medical trauma related sequelae
Medical Sequelae in COVID-19 Survivors | Screening-Month 36
  Characterize the medical sequelae and persistent symptoms following recovery from COVID-19 in a cohort of disease survivors.
Incidence of reinfection with COVID-19 | Screening-Month 36
  Evaluate survivors for evidence of re-infection with future waves of COVID-19 to determine if initial infection confers long-term protective immunity
Incidence of clinical silent infection | Screening-Month 36
  Determine the incidence of clinically silent infection in household contacts
Antibody and cell-mediated immune responses to SARS-CoV-2 over time | Screening-Month 36
  Characterize evolution of the antibody and T cell-mediated responses to SARS-CoV-2 in survivors over time
Antibody and cell-mediated immune responses to SARS-CoV-2 | Screening-Month 36
  Characterize antibody and cell-mediated immune responses to SARS-CoV-2 in disease survivors

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Sneller, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sneller MC, Liang CJ, Marques AR, Chung JY, Shanbhag SM, Fontana JR, Raza H, Okeke O, Dewar RL, Higgins BP, Tolstenko K, Kwan RW, Gittens KR, Seamon CA, McCormack G, Shaw JS, Okpali GM, Law M, Trihemasava K, Kennedy BD, Shi V, Justement JS, Buckner CM, Blazkova J, Moir S, Chun TW, Lane HC. A Longitudinal Study of COVID-19 Sequelae and Immunity: Baseline Findings. Ann Intern Med. 2022 Jul;175(7):969-979. doi: 10.7326/M21-4905. Epub 2022 May 24. PMID 35605238
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-I-0123.html